CLINICAL TRIAL: NCT06866860
Title: Evaluation of Internally Irrigated and Externally Irrigated Surgical Guide Design for Placement of Dental Endosseous Implants in Mandibular Posterior Region (Randomized Controlled Clinical Trial)
Brief Title: Internally Irrigated and Externally Irrigated Surgical Guide Design for Placement of Dental Endosseous Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant Lecturer of Dental Public Health and biostatistical consultanat, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0810-12/2023
Record Dates: First submitted 2025-03-02; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Dental Implant

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental)
  Interventions: Other: Implant surgical guide with internal irrigation
- Control group (Active Comparator)
  Interventions: Other: Conventional implant surgical guide with external irrigation

INTERVENTIONS:
Other: Implant surgical guide with internal irrigation — * Virtual surgical plan will be completed in the implant planning software (BlueSky plan, BlueSky Bio, USA), and the implant type, position, and sleeve height will be adjusted.
  * The entry point of the surgical drill into the alveolar bone will be identified.
  * An irrigation channel will be added, directed toward the entry point of the drill and adjusted to have the same diameter as the irrigation system tube.
  Arms: Study group
Other: Conventional implant surgical guide with external irrigation — Virtual surgical plan will be completed in the implant planning software (BlueSky plan, BlueSky Bio, USA), and the implant type, position, and sleeve height will be adjusted. Conventional guide will be printed
  Arms: Control group

SUMMARY:
Background: Patient specific surgical guides (PSG) have been widely used to achieve a precise 3D implant position. However, they prevent external cooling systems from reaching the osteotomy site sufficiently. So, heat generated during guided implant surgery is greater than free hand technique. Adding internal irrigation channel to the conventional surgical guides allows better diffusion of irrigation to the osteotomy site and reduces heat generation.

Aim of the study: Is to introduce a patient specific surgical guide design with internal irrigation system and compare it to the conventional surgical guide with external irrigation clinically through bone temperature, implant stability and radiographically by CBCT through crestal bone loss and bone density.

ELIGIBILITY:
Inclusion Criteria:

* Patient with missing mandibular posterior premolar or molar teeth.
* Tooth extraction at the implant sites was performed at least 4 months before the surgery.
* Residual alveolar bone height more than 10 mm.
* With minimum alveolar bucco-lingual dimension of 6 mm.
* Free from any systemic disease or local pathological lesions that may affect bone healing or contraindicate implant placement.

Exclusion Criteria:

* Severe atrophic alveolar ridge (height less than 10mm, width less than 6mm).
* Bad oral hygiene ( Silness-Löe index (score 2-3).
* Heavy smoker (smoke greater than or equal 25 cigarettes per day).
* Presence of acute infections or periapical lesions in adjacent teeth.
* Parafunctional habits.
* Pregnant females.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2024-04-04 (Actual); Primary Completion 2024-10-17 (Actual); Study Completion 2024-10-17 (Actual)

PRIMARY OUTCOMES:
change in implant stability | Baseline and 4 months
  Osstell will be used to objectively and non-invasively determine implant stability and to assess the progress of osseointegration without jeopardizing the healing process.
  This method is based on determining whether or not an implant is stable enough. The result is presented as an ISQ value of 1-100. The higher the ISQ, the more stable the implant
change in postoperative oedema | 2nd day, 1 week and 2 weeks
  This will be measured as follows:
  None (no inflammation). Mild (intraoral swelling confined to the surgical field). Moderate (extraoral swelling in the surgical zone). Severe (extraoral swelling spreading beyond the surgical zone).

SECONDARY OUTCOMES:
Presence of intra or postoperative complications | 4 months
  Bone overheating. Bone fenestration. Wound dehiscence. Peri-implantitis.
change in crestal bone loss | baseline and 4 months
  A CBCT was obtained immediately post operatively T1 and after 4 months T2 and evaluated using (BlueSky plan, BlueSky Bio, USA) to asses Crestal bone loss.
change in bone density | baseline and 4 months
  A CBCT was obtained immediately post operatively T1 and after 4 months T2 and evaluated using (BlueSky plan, BlueSky Bio, USA) to asses Bone density using Hounsfield Unit (HU).

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Clinic of Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Alexandria University, Egypt, Alexandria, Azarita, Egypt